CLINICAL TRIAL: NCT00104520
Title: A Phase 3, Double-Blind, Multicenter, Randomized, Placebo-Controlled Trial With Aztreonam Lysinate for Inhalation in Cystic Fibrosis Patients With Pulmonary P. Aeruginosa Requiring Frequent Antibiotics (AIR-CF2)
Brief Title: Safety and Efficacy Study of Aztreonam for Inhalation Solution (AZLI) in Cystic Fibrosis Patients With P. Aeruginosa
Acronym: AIR-CF2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Mark Bresnik, MD, Director, Clinical Research, Gilead Sciences, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-AI-005
Record Dates: First submitted 2005-03-01; First posted 2005-03-02 (Estimated); Results first posted 2011-03-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2010-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Pseudomonas aeruginosa; Pulmonary Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (pooled two times a day [BID]/three times a day [TID]) (Placebo Comparator)
  Interventions: Drug: Placebo two times a day (BID)/three times a day (TID)
- AZLI (pooled two times a day [BID]/three times a day [TID]) (Experimental)
  Interventions: Drug: AZLI 75 mg two times a day (BID)/three times a day (TID)

INTERVENTIONS:
Drug: AZLI 75 mg two times a day (BID)/three times a day (TID)
  Arms: AZLI (pooled two times a day [BID]/three times a day [TID])
Drug: Placebo two times a day (BID)/three times a day (TID)
  Arms: Placebo (pooled two times a day [BID]/three times a day [TID])

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of aztreonam for inhalation solution (AZLI) in patients with cystic fibrosis (CF) and lung infection due to Pseudomonas aeruginosa (PA).

DETAILED DESCRIPTION:
Patients with CF often have lung infections that occur repeatedly or worsen over time. The lung infections are often caused by a bacteria called PA. Treatment with antibiotics can stop or slow down the growth of the bacteria. The antibiotics may be given by mouth, intravenously (IV), or by inhalation as a mist. The purpose of this study was to evaluate the safety and efficacy of aztreonam for inhalation solution (AZLI), an investigational formulation of the antibiotic administered using the eFlow® Electronic Nebulizer by PARI GmbH, in CF patients with PA.

In this study, participants were screened for eligibility at Visit 1 (Day -42) and returned to the center for Visit 2 after a 14-day evaluation period. At Visit 2 (Day -28), participants began a 28-day course of open-label Tobramycin Inhalation Solution (TIS). At Visit 3 (Day 0), following completion of the 28-day course of TIS, participants began randomized, blinded treatment with either AZLI twice a day (BID) or three times a day (TID) or placebo BID or TID, and continued treatment for a total of 28 days, with a clinic visit at Day 14 (Visit 4) and at the end of treatment (Visit 5 [Day 28]). Participants returned for visits every 2 weeks for 8 weeks after the end of the blinded treatment (Visits 6 to 9 [Days 42 to 84]).

Two hundred and forty-seven participants were treated in the TIS phase of this study. Two hundred and eleven subjects completed the TIS phase and were treated in the placebo-controlled phase with study drug (AZLI or placebo).

ELIGIBILITY:
Inclusion Criteria:

* CF as diagnosed by:

  1. Documented sweat chloride greater than or equal to 60 mEq/L by quantitative pilocarpine iontophoresis test; or
  2. Two well-characterized genetic mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene; or
  3. Abnormal nasal potential difference with accompanying symptoms characteristic of CF.
* PA present in expectorated sputum or throat swab culture at Screening.
* Participants must have received three or more courses of TIS within the previous 12 months.
* Participants on chronic azithromycin must have had no change in regimen in the previous 3 months and must have had a need for TIS and/or additional antipseudomonal therapy since initiation of azithromycin.
* Forced expiratory volume in 1 second (FEV1) between (and including) 25% and 75% predicted at Screening.
* Ability to perform reproducible pulmonary function tests.
* Arterial oxygen saturation (SaO2) greater than or equal to 90% on room air at Screening.

Exclusion Criteria:

* Current use of oral corticosteroids in doses exceeding the equivalent of 10 mg prednisone a day or 20 mg prednisone every other day.
* History of sputum or throat culture swab yielding Burkholderia cepacia in the past 2 years.
* History of daily continuous oxygen supplementation or requirement for more than 2 liters/minute at night.
* Administration of any investigational drug or device within 28 days of Screening (Visit 1) or within 6 half-lives of the investigational drug (whichever was longer).
* Known local or systemic hypersensitivity to monobactam antibiotics.
* Inability to tolerate inhalation of a short acting Beta-2 agonist.
* Changes in antimicrobial, bronchodilator, anti-inflammatory, or corticosteroid medications within 7 days before Screening or between Screening and the next visit.
* Changes in physiotherapy technique or schedule within 7 days before Screening or between Screening and the next visit.
* History of lung transplantation.
* A chest X-ray indicating abnormal findings at Screening or within the previous 90 days.
* Abnormal renal or hepatic function or serum chemistry at Screening (aspartate aminotransferase [AST], alanine aminotransferase [ALT] greater than 5 times the upper limit of normal range; Creatinine greater than 2 times the upper limit of normal range).
* Positive pregnancy test at Screening.
* Female of childbearing potential who was lactating or in the opinion of the investigator was not practicing acceptable birth control.
* Any serious or active medical or psychiatric illness, which in the opinion of the investigator would have interfered with participant treatment, assessment, or compliance with the protocol.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2005-02; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen McCoy, MD, Principal Investigator — Nationwide Children's Hospital
Locations (56):
- United States (56):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, San Diego, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Medical Care Program, Oakland, California
  - Children's Hospital, Orange Co., Orange, California
  - Stanford University Hospital and Medical Center, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - Children's Hospital, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - University of Florida Health Sciences Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Jacksonville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - Pediatric Pulmonary Associates, Florida, St. Petersburg, Florida
  - Emory Healthcare, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Children's Memorial Hospital/Northwestern University, Chicago, Illinois
  - Chicago Children's Asthma Respiratory and Exercise Specialists, Glenview, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - North Suburban Pulmonary / Critical Care Consultants, Niles, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Maine Medical Center, Portland, Maine
  - Children's Hospital, Boston, Boston, Massachusetts
  - Floating Hospital for Children, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan/Wayne State University, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Lung Specialists, Ltd., Las Vegas, Nevada
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Albany Medical College, Albany, New York
  - Long Island College Hospital, Brooklyn, New York
  - Children's Hospital of Buffalo, Buffalo, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - State University of New York Stony Brook, Stony Brook, New York
  - Children's Hospital of Westchester Medical Center/New York Medical College, Valhalla, New York
  - Akron Children's Hospital, Akron, Ohio
  - Columbus Children's Hospital, Ohio State University, Columbus, Ohio
  - Children's Medical Center, Dayton, Ohio
  - Dr. Santiago Reyes, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Penn State University Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburg, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Pediatric Pulmonary Associates, South Carolina, Columbia, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Alamo Clinical Research Associates, San Antonio, Texas
  - Pediatric Pulmonary Center, Richmond, Virginia
  - Children's Hospital and Regional Medical Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Derived] Quittner AL, Modi AC, Wainwright C, Otto K, Kirihara J, Montgomery AB. Determination of the minimal clinically important difference scores for the Cystic Fibrosis Questionnaire-Revised respiratory symptom scale in two populations of patients with cystic fibrosis and chronic Pseudomonas aeruginosa airway infection. Chest. 2009 Jun;135(6):1610-1618. doi: 10.1378/chest.08-1190. Epub 2009 May 15. PMID 19447923
- [Derived] McCoy KS, Quittner AL, Oermann CM, Gibson RL, Retsch-Bogart GZ, Montgomery AB. Inhaled aztreonam lysine for chronic airway Pseudomonas aeruginosa in cystic fibrosis. Am J Respir Crit Care Med. 2008 Nov 1;178(9):921-8. doi: 10.1164/rccm.200712-1804OC. Epub 2008 Jul 24. PMID 18658109

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 56 sites in the United States. Date of first enrollment was 24 February 2005, and date of last participant follow-up was 07 September 2006.
Pre-assignment Details: Subjects were randomized in 1:1:2:2 ratio to placebo twice a day (BID) or three times a day (TID) and AZLI BID or TID, respectively. A total of 211 subjects were included in the ITT analyses: 38 placebo BID, 38 placebo TID, 69 AZLI BID, and 66 AZLI TID. All analyses were conducted on pooled placebo (n = 76) versus pooled AZLI (n = 135) groups.
Groups:
- Placebo (Pooled BID/TID): Placebo (5 mg/mL lactose when reconstituted in diluent [0.17% saline]; sterile, pH 4.2 to 7.5, and osmolality 200 to 400 mOsmol/kg). Placebo was self-administered twice daily (BID) or three times daily (TID) by inhalation using the investigational nebulizer. All analyses were conducted on the pooled placebo vs pooled AZLI treatment groups.
- AZLI (Pooled BID/TID): AZLI (75 mg/mL aztreonam lysine when reconstituted in diluent [0.17% saline]; sterile, pH 4.2 to 7.0, and osmolality 300 to 550 mOsmol/kg). AZLI was self-administered by inhalation BID or TID using the investigational nebulizer. All analyses were conducted on the pooled placebo vs pooled AZLI treatment groups.
Period: Overall Study
Arm/Group | Placebo (Pooled BID/TID) | AZLI (Pooled BID/TID)
Started | 76 | 135
Completed | 26 | 64
Not Completed | 50 | 71
Not completed — Unrelated adverse event | 34 | 47
Not completed — Study drug intolerance | 0 | 1
Not completed — Related adverse event | 13 | 15
Not completed — Lost to Follow-up | 1 | 0
Not completed — Noncompliance | 0 | 2
Not completed — Personal/administrative | 1 | 1
Not completed — Other | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Pooled BID/TID) | AZLI (Pooled BID/TID) | Total
Number analyzed (Participants) | 76 | 135 | 211
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 34 | 46
  Between 18 and 65 years | 63 | 101 | 164
  >=65 years | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 27.9 (10.4) | 25.3 (10.2) | 26.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 59 | 90
  Male | 45 | 76 | 121
Region of Enrollment [Number; unit: participants]
  United States | 76 | 135 | 211

OUTCOME MEASURES:

1. Primary Outcome: Time to Need for Inhaled or Intravenous (IV) Antipseudomonal Antibiotics
Description: The primary endpoint was time to need for a course of inhaled or IV antipseudomonal antibiotics with documented physician assessment of need for antibiotics. Antipseudomonal Antibiotic need was documented based on the presence of at least one of the following four symptoms predictive of pulmonary exacerbation: decreased exercise tolerance, increased cough, increased sputum / chest congestion, decreased appetite, or other.
Time Frame: Day 0 to Day 84 (end of study)
Population: Analysis based on intents to treat (ITT) population (all participants randomized to treatment who received at least part of one dose of study drug).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo (Pooled BID/TID) | AZLI (Pooled BID/TID)
Number analyzed (Participants) | 76 | 135
Days | 71 [57 to 97] | 92 [89 to NA] — NA = not estimable
Statistical Analysis 1: Comparison: Placebo (Pooled BID/TID) vs AZLI (Pooled BID/TID); H0: no difference between AZLI and placebo (pooled treatment groups) in time to need for inhaled or IV antibiotics. Assuming 2-sided significance level of 0.05, ~210 subjects (70 in each AZLI group, 35 in each placebo group) provided >90% power to reject null hypothesis based on Lakatos normal approximation method with weights being one. Therefore, 250 subjects were to be randomized at Visit 2 (Day -28) to ensure at least 210 participants entered double-blind treatment period at Day 0; Test type: Superiority or Other; p = 0.0070, Log Rank — Analysis based on 2-sided test with 0.05 a priori threshold for statistical significance. No adjustments were made for multiple comparisons

2. Secondary Outcome: Change in Cystic Fibrosis Questionnaire - Revised (CFQ-R) Respiratory Symptoms Scale (RSS) Score
Description: The CFQ-R was administered at Day -28, baseline, Day 14, Day 28, and Day 84 (end of study). The endpoint was change in respiratory symptoms from baseline, assessed with the CFQ-R RSS (range of scores [units]: 0-100; higher scores indicate fewer symptoms).
Time Frame: Day 0 to Day 28
Population: Analysis based on ITT population (all participants randomized to tx who received at least part of one dose of study drug). Missing baseline data were not imputed. Missing post-baseline data were imputed using worst-case value for participants who withdrew due to AE or study drug intolerance. For all other missing data, LOCF method was used.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo (Pooled BID/TID) | AZLI (Pooled BID/TID)
Number analyzed (Participants) | 73 | 132
Units on a scale | -0.66 (1.708) | 4.34 (1.27)
Statistical Analysis 1: Comparison: Placebo (Pooled BID/TID) vs AZLI (Pooled BID/TID); Null hypothesis was there is no difference between 75 mg AZLI and placebo (pooled treatment groups) in change from baseline in CFQ-R RSS scores; Test type: Superiority or Other; p = 0.0196, ANCOVA — No adjustments were made for multiple comparisons; ANCOVA model included terms for treatment and baseline value; Mean Difference (Final Values) = 5.01, 95% CI 2-sided [0.81 to 9.21]

3. Secondary Outcome: Percent Change in Forced Expiratory Volume in 1 Second (FEV1) (L)
Description: Spirometry was performed at each visit. FEV1 was recorded according to American Thoracic Society (ATS) guidelines.
  FEV1(L) is the measurement of the volume of air (expressed in liters) exhaled in 1 second.
  The percent change in this parameter from Day 0 to Day 28 was determined for each treatment group.
Time Frame: Day 0 to Day 28
Population: Analysis based on ITT population (all participants who received at least part of one dose of study drug). Missing baseline data were not imputed. Missing post-baseline data were imputed using worst-case value for participants who withdrew due to an AE or study drug intolerance. For all other missing data, LOCF imputation method was used.
Measure: Least Squares Mean (Standard Error); unit: Percent change in FEV1 (L)
Arm/Group | Placebo (Pooled BID/TID) | AZLI (Pooled BID/TID)
Number analyzed (Participants) | 76 | 135
Percent change in FEV1 (L) | -2.363 (1.534) | 3.917 (1.151)
Statistical Analysis 1: Comparison: Placebo (Pooled BID/TID) vs AZLI (Pooled BID/TID); Null hypothesis was there is no difference between 75 mg AZLI and placebo (pooled treatment groups) in percent change from baseline in FEV1 (L); Test type: Superiority or Other; p = 0.0012, ANCOVA — No adjustments were made for multiple comparisons; ANCOVA model included terms for treatment and baseline value; Mean Difference (Final Values) = 6.280, 95% CI 2-sided [2.500 to 10.060]

4. Secondary Outcome: Number of Hospitalization Days
Description: Details of all hospitalizations, including the dates of admission and discharge, were recorded on the electronic case report form (eCRF).
Time Frame: Day 0 to Day 84
Population: Analysis based on ITT population (all participants randomized to treatment who received at least part of one dose of study drug). No imputation methods were used for the analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo (Pooled BID/TID) | AZLI (Pooled BID/TID)
Number analyzed (Participants) | 76 | 135
Days | 0.5 (2.4) | 0.9 (3.9)

5. Secondary Outcome: Change From Baseline in Pseudomonas Aeruginosa (PA) Log10 Colony Forming Units (CFU) Per Gram of Sputum
Description: Sputum samples were collected at all participant visits of the study for analysis of microbiology endpoints. Sputum samples were processed for qualitative and quantitative culture of PA (each morphotype). Due to the skewness of the distribution of CFU data, the data were transformed using the base 10 logarithm, in an attempt to normalize the data and allow for parametric tests, before calculating changes. To account for zero values, 1 was added to each CFU measurement before being transformed. Any CFU data values where PA was not isolated from a valid culture were set to zero.
Time Frame: Day 0 to Day 28
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Log10 PA CFUs/gram of sputum
Arm/Group | Placebo (Pooled BID/TID) | AZLI (Pooled BID/TID)
Number analyzed (Participants) | 57 | 95
Log10 PA CFUs/gram of sputum | 0.225 (0.209) | -0.434 (0.167)
Statistical Analysis 1: Comparison: Placebo (Pooled BID/TID) vs AZLI (Pooled BID/TID); Null hypothesis was there is no difference between 75 mg AZLI and placebo (pooled treatment groups) in mean change from baseline in log10 PA CFUs in sputum; Test type: Superiority or Other; p = 0.0059, ANCOVA; ANCOVA model included terms for treatment and baseline highest MIC of aztreonam for PA (<=2, 4-8, 16-128 or >=256 μg/mL) value; Mean Difference (Final Values) = -0.659, 95% CI 2-sided [-1.125 to -0.193]

6. Other Pre Specified Outcome: Number of Participants With Other Pathogens
Description: Sputum samples were collected at all visits for quantitative and qualitative culture for Staphylococcus aureus, Burkholderia cepacia, Stenotrophomonas maltophilia, and Achromobacter xylosoxidans.
  Number of participants with other pathogens at baseline and at the end of treatment (28 days) are reported.
Time Frame: Day 0 and Day 28
Population: Analysis based on ITT population (all participants who received at least part of one dose of study drug). No imputation methods were used for the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo (Pooled BID/TID) | AZLI (Pooled BID/TID)
Number analyzed (Participants) | 76 | 135
Participants
  S. aureus - Day 0 | 23 | 58
  S. aureus - Day 28 | 23 | 63
  B. cepacia - Day 0 | 0 | 0
  B. cepacia - Day 28 | 0 | 0
  S. maltophilia - Day 0 | 9 | 18
  S. maltophilia - Day 28 | 8 | 19
  A. xylosoxidans - Day 0 | 6 | 10
  A. xylosoxidans - Day 28 | 6 | 7

7. Other Pre Specified Outcome: Minimum Concentration of Aztreonam Inhibiting 50% (MIC50) and 90% (MIC90) of All PA Isolates (μg/mL)
Description: The aztreonam susceptibility of PA isolates from sputum samples (collected at all visits) was assessed.
  MIC50 = minimum inhibitory concentration (minimum concentration of an agent that inhibits 50% of isolates from a particular organism).
  MIC90 = minimum inhibitory concentration (minimum concentration of an agent that inhibits 90% of isolates from a particular organism).
  MIC50 and MIC90 values are single measurements for the entire population and not measured on a per-participant basis.
Time Frame: Day 0 to Day 28
Population: as for outcome 6
Measure: Number; unit: μg/mL
Arm/Group | Placebo (Pooled BID/TID) | AZLI (Pooled BID/TID)
Number analyzed (Participants) | 76 | 135
μg/mL
  Baseline MIC50 | 1 | 2
  Day 28 MIC50 | 1 | 4
  Baseline MIC90 | 64 | 32
  Day 28 MIC90 | 64 | 64

ADVERSE EVENTS:
Time Frame: AEs that first occurred or worsened after the first dose of study drug through 30 days after the last dose (Day 0 to Day 56) are summarized.
Description: An AE was any physical or clinical worsening in symptoms or disease (including clinically significant change in lab values) experienced by participant at any time during treatment period of study, whether or not event was considered related to study participation or procedures. Participants were only counted once within an SOC and preferred term.
Arm/Group | Placebo (Pooled BID/TID) | AZLI (Pooled BID/TID)
Serious Adverse Events (participants affected / at risk) | 3/76 | 13/135
Other Adverse Events (participants affected / at risk) | 65/76 | 121/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Pooled BID/TID) (N=76) | AZLI (Pooled BID/TID) (N=135)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest X-ray abnormal (Investigations) | 0 (0) | 1 (1)
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Exercise tolerance decreased (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Forced expiratory volume decreased (Investigations) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neurological symptoms (Nervous system disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Pulmonary function test decreased (Investigations) | 0 (0) | 4 (4)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Pooled BID/TID) (N=76) | AZLI (Pooled BID/TID) (N=135)
Abdominal pain (Gastrointestinal disorders) | 2 | 10
Abdominal pain upper (Gastrointestinal disorders) | 3 | 7
Blood glucose increased (Investigations) | 4 | 2
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 6 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 51 | 81
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 10 | 11
Decreased appetite (Metabolism and nutrition disorders) | 11 | 11
Diarrhoea (Gastrointestinal disorders) | 1 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Exercise tolerance decreased (General disorders) | 10 | 11
Fatigue (General disorders) | 12 | 14
Forced expiratory volume decreased (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 14 | 17
Headache (Nervous system disorders) | 9 | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 28
Nausea (Gastrointestinal disorders) | 4 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 18
Productive cough (Respiratory, thoracic and mediastinal disorders) | 27 | 49
Pulmonary function test decreased (Investigations) | 8 | 9
Pyrexia (General disorders) | 2 | 16
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 15 | 20
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 14
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Sinus headache (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Vomiting (Gastrointestinal disorders) | 5 | 9
Wheezing (Respiratory, thoracic and mediastinal disorders) | 9 | 22

LIMITATIONS AND CAVEATS:
The study was designed such that participants were discontinued from study participation upon meeting the primary endpoint (time to need for inhaled or IV antipseudomonal antibiotics).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and investigator may publish or present the results of the trial generated there with prior written consent of Gilead; or 2 years after the trial has ended at all institutions. Proposed publications/target venue must go to Gilead 30 days (manuscripts) or 15 days (abstracts/presentations) prior. Any Gilead confidential information in the document(s) must be deleted, or if requested publication delayed for up to 45 days to permit Gilead to obtain intellectual property protection.